CLINICAL TRIAL: NCT02058394
Title: Postoperative Events in Patients With and Without Retained Nuclear Fragments in the Anterior Vitreous After Routine Phacoemulsification
Brief Title: Retained Lens Fragments After Phacoemulsification
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ophthalmic Consultants, Corneal and Refractive Surgery Associates, PC (Other)
Responsible Party: Principal Investigator, David Ritterband, MD, Ophthalmic Consultants, Corneal and Refractive Surgery Associates, PC
Other Study IDs: 12.08
Record Dates: First submitted 2014-02-04; First posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Cataract
Keywords: Retained nuclear lens fragments; Phacoemulsification; Cataract Surgery
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cataract Phacoemulsification: Subjects will be recruited serially from eligible candidates on the basis of presentation for cataract evaluation and subsequent cataract surgery with phacoemulsification.
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — Subjects will be recruited serially from eligible candidates on the basis of presentation for cataract evaluation and subsequent cataract surgery with phacoemulsification.

SUMMARY:
The purpose of this study is to investigate postoperative events in patients noted to have retained nuclear fragments in the anterior vitreous during routine phacoemulsification and in those who did not.

DETAILED DESCRIPTION:
In this study, we investigate whether presence of retained nuclear fragments in the anterior vitreous noted during uncomplicated cataract surgery is associated with higher incidence of postoperative adverse events. We will be assessing events including cystoid macular edema, iritis, elevated intraocular pressure, and retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* Routine cataract surgery with phacoemulsification

Exclusion Criteria:

* Pre-existing macular edema
* Active uveitis
* Intraocular exclusion surgeries
* Significant ocular trauma
* Evidence of phacodonesis or zonular weakness .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited serially from eligible candidates on the basis of presentation for cataract evaluation and subsequent cataract surgery with phacoemulsification.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Macular edema | 1 month postoperatively
  Proportion of eyes with clinical macular edema and subclinical macular edemas measured by OCT at 1 month postoperatively

SECONDARY OUTCOMES:
Intraocular inflammation | 1 month postoperativley
  Proportion of eyes with persistent anterior chamber inflammation requiring medical treatment at 1 month postoperatively
Elevated intraocular pressure | 1 month postoperatively
  Proportion of eyes with intraocular pressure increase requiring medical or surgery treatment at 1 month postoperatively
Macular Edema | 1 week postoperatively
  Proportion of eyes with clinical macular edema and subclinical macular edemas measured by OCT at 1 week postoperatively
Intraocular Inflammation | 1 week postoperatively
  Proportion of eyes with persistent anterior chamber inflammation requiring medical treatment at 1 week postoperatively
Elevated Intraocular Pressure | 1 week postoperatively
  Proportion of eyes with intraocular pressure increase requiring medical or surgery treatment at 1 week postoperatively
Macular Edema | 3 months postoperatively
  Proportion of eyes with clinical macular edema and subclinical macular edemas measured by OCT at 3 months postoperatively
Intraocular Inflammation | 3 months
  Proportion of eyes with persistent anterior chamber inflammation requiring medical treatment at 3 months postoperatively

OTHER OUTCOMES:
Surgical Complications | Intraoperatively
  Proportion of eyes with surgical adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: David Ritterband, MD, Principal Investigator — Ophthalmic Consultants, Cornea and Refractive Surgery Assoicates, PC
Locations (1):
- Ophthalmic Consultants, Corneal and Refractive Surgery Associates, PC, New York, New York, United States